CLINICAL TRIAL: NCT05348460
Title: Effects of a Single Oral Dose of KETone Ester ON Exercise Performance in Patients With Chronic Heart Failure
Acronym: KETONE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201900710
Record Dates: First submitted 2022-03-04; First posted 2022-04-27 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Heart Failure
Keywords: Heart Failure; Ketone Body; HFrEF; Skeletal Muscle Metabolism; Mitochondrial Ketone Oxidation; 31P MRS; Pi/Pcr
MeSH Terms: conditions — Heart Failure | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled cross-over design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone - Placebo treatment (Other): Patients will first receive a supplemental drink containing a ketone ester before performing the 31P MRS exercise protocol. After 1-2 weeks, subjects will cross-over and repeat the 31P MRS exercise protocol, this time after receiving the placebo treatment.
  Interventions: Dietary Supplement: Ketone ester drink (DeltaG®, 500 mg/kg body weight); Dietary Supplement: Taste-matched, isovolumic placebo drink
- Placebo - Ketone treatment (Other): Patients will first receive a placebodrink before performing the 31P MRS exercise protocol. After 1-2 weeks, subjects will cross-over and repeat the 31P MRS exercise protocol, this time after receiving the supplemental drink containing a ketone ester.
  Interventions: Dietary Supplement: Ketone ester drink (DeltaG®, 500 mg/kg body weight); Dietary Supplement: Taste-matched, isovolumic placebo drink

INTERVENTIONS:
Dietary Supplement: Ketone ester drink (DeltaG®, 500 mg/kg body weight) — In a double blind fashion, subjects will receive a ketone ester drink ór a taste-matched, isovolumic placebo drink and will then perform the 31P MRS exercise protocol. After 1-2 weeks, subjects will cross-over and repeat the 31P MRS exercise protocol, this time receiving the other treatment.
Dietary Supplement: Taste-matched, isovolumic placebo drink — In a double blind fashion, subjects will receive a ketone ester drink ór a taste-matched, isovolumic placebo drink and will then perform the 31P MRS exercise protocol. After 1-2 weeks, subjects will cross-over and repeat the 31P MRS exercise protocol, this time receiving the other treatment.

SUMMARY:
In a randomized, double-blind, placebo-controlled cross-over design, subjects will either receive a supplemental drink containing a commercially available ketone ester (DeltaG®, 500 mg/kg body weight), or a taste matched, isovolumic placebodrink and will then perform the 31phosphorus Magnetic Resonance Spectroscopy (31P MRS) exercise protocol. After 1-2 weeks, subjects will cross-over and repeat the 31P MRS exercise protocol, this time receiving the other treatment.

DETAILED DESCRIPTION:
The goal of this study is to investigate if oral ketone supplementation stimulates mitochondrial ATP production and improves exercise performance in patients with chronic HF. In a randomized, double-blind, placebo-controlled cross-over design, subjects will either receive a supplemental drink containing a commercially available ketone ester (DeltaG®, 500 mg/kg body weight), or a taste matched, isovolumic placebodrink and will then perform the 31P MRS exercise protocol. After 1-2 weeks, subjects will cross-over and repeat the 31P MRS exercise protocol, this time receiving the other treatment. Endpoints include rate and magnitude of change in phosphocreatine (PCr) and inorganic phosphate (Pi) concentrations from baseline to maximum exercise, rate and magnitude of change in PCr and Pi concentrations during recovery, rates and magnitude of change in intramuscular pH during exercise and recovery, maximal exercise performance and change in concentrations of beta-hydroxybutyrate and other metabolites before consumption of the supplemental drink, after consumption of the supplemental drink and after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Heart Failure NYHA II - III
* LVEF ≤40%
* Stable for the last 1 month prior to the study

Exclusion Criteria:

* Age <18 years;
* Unable or unwilling to undergo exercise MRI (physical disabilities, claustrophobia);
* Unable to complete the exercise protocol during the screening visit according to the professional opinion of the investigators;
* Comorbidities which can influence study results such as muscular dystrophies, peripheral artery disease, diabetes mellitus, severe anaemia (defined as Hb ≤6 mmol/L);
* Pregnant/trying to get pregnant/breastfeeding during the period from the first exercise test until 4 weeks after the last exercise test);
* Absolute contra-indications to undergo MRI according to the current UMCG protocols and guidelines (e.g. non-conditional medical device, recent device implantation, incompatible ferromagnetic objects in the body).
* BMI < 16 kg/m2; BMI > 35 kg/m2
* Unable to understand study procedures;
* Unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Phosphocreatine (PCr) and inorganic phosphate (Pi) concentrations from baseline to maximum exercise | During study-visit
  Rate and magnitude of change in PCr and Pi concentrations from baseline to maximum exercise.

SECONDARY OUTCOMES:
Rate and magnitude of change in PCr and Pi concentrations during recovery | During study visit
  Rate and magnitude of change in PCr and Pi concentrations during recovery of change in PCr and Pi is expressed as change in Pi/PCr (ΔPi/PCr)
Intramuscular pH | During study visit
  Rates and magnitude of change in intramuscular pH during exercise and recovery
Maximal exercise performance | During study visit
  Maximal exercise performance
Change in concentrations of beta-hydroxybutyrate and other metabolites before consumption of the supplemental drink, after consumption of the supplemental drink and after exercise | During study visit
  Change in concentrations of beta-hydroxybutyrate and other metabolites before consumption of the supplemental drink, after consumption of the supplemental drink and after exercise

CONTACTS AND LOCATIONS:
Overall Officials: Daan Westenbrink, MD PhD, Principal Investigator — Unversity Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands